CLINICAL TRIAL: NCT01865032
Title: Pivotal Trials: Evaluation of a Rapid Diagnostic Device, CL Detect™ Rapid Test, for the Diagnosis of Cutaneous Leishmaniasis in the United States
Brief Title: Evaluation of CL Detect™ Rapid Test to Detect Cutaneous Leishmaniasis
Status: Completed | Type: Observational
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Collaborators: InBios International, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: S-12-19
Record Dates: First submitted 2013-05-23; First posted 2013-05-30 (Estimated); Last update posted 2014-09-08 (Estimated); Status verified 2014-09

CONDITIONS: Skin Diseases
MeSH Terms: conditions — Skin Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — dental broach samples in lysis buffer
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Skin Ulcers: Skin ulcers. No intervention. Subjects will be followed up by their respective primary providers.

SUMMARY:
This study is a single-site trial assessing the specificity of CL Detect™ Rapid Test versus the gold standard for Leishmania diagnosis in the US which is microscopic identification of Leishmania amastigotes in a stained lesion sample. Subjects will be patients who present for dermatology consultation with a primarily ulcerated lesion. After informed consent is obtained and the subject is screened for eligibility, 2 diagnostic samples will be collected from the subject's lesion in the following order: 1) one sample will be obtained with a dental broach for use with the CL Detect™ Rapid Test and 2) a second sample will be obtained by scraping for use in the microscopic identification of amastigotes. Samples will be analyzed by microscopy and CL Detect™ Rapid Test. The CL Detect™ Rapid Test will be performed by different operators who are clinical staff members. These staff members, blinded to each other's results, will evaluate the samples from each method independently. Each of the 150 study subjects will be followed administratively to the point where a diagnosis is established (if possible) for their tested lesion, even if that diagnosis is not cutaneous leishmaniasis (CL). If a specific diagnosis cannot be determined for a non-CL lesion, the investigator will assign a "likely etiology" (eg, infectious, oncological, immunological, vascular, or "undetermined/other" origin). Based on the diagnosis determined for each lesion, subjects will be referred for appropriate treatment.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Subject is able to give written informed consent
* Subject has a skin ulcer that satisfies the following criteria for an index lesion:
* less than 4 months in age
* primarily ulcerative, not purely verrucous or nodular, and does not have clear clinical evidence of cellulitis
* in a location suitable for collecting samples by dental broach and scraping
* In the opinion of the investigator, the subject is capable of understanding and complying with the protocol

Exclusion Criteria:

* Received treatment for leishmaniasis or any treatment to the lesion even if not previously diagnosed as leishmaniasis such as azoles, cryotherapy, imiquimod, thermotherapy, photodynamic therapy, within 2 months prior to signing the consent form, with the exception of mercurochrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Dermatology clinic
Sampling Method: Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2013-06; Primary Completion 2013-08 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Specificity | 1 hour
  Specificity will be presented for the CL Detect™ Rapid Test device against the reference method (microscopy). Specificity will be calculated as the number of true negatives divided by the sum of the number of true negatives plus the number of false positives times 100%.

SECONDARY OUTCOMES:
False positive rate | 1 hour
  α, type 1 error, calculated as 1-specificity times 100%
False negative rate | 1 hour
  β, type 2 error, calculated as 1-sensitivity times 100%

CONTACTS AND LOCATIONS:
Overall Officials: Mark Lebwohl, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Mount Sinai School of Medicine, New York, New York, United States